CLINICAL TRIAL: NCT00571818
Title: The Prospective Evaluation of Pancreatic Function in Pancreas Transplant Recipients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Diagnostic
Other Study IDs: 0114-00-FB
Record Dates: First submitted 2007-12-11; First posted 2007-12-12 (Estimated); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Transplant; Diabetes
Keywords: euglycemic; transplant; pancreas; hyperglycemic; kidney
MeSH Terms: conditions — Diabetes Mellitus | interventions — Glucose Tolerance Test

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Euglycemic pancreas transplant recipients (Active Comparator): Participants receiving a pancreas transplant who have blood glucose level is within the normal range
  Interventions: Procedure: Oral glucose tolerance test; Procedure: IV Glucose Tolerance Test
- Hyperglycemic pancreas transplant recipients (Active Comparator): Participants receiving a pancreas transplant who have high blood glucose (blood sugar)
  Interventions: Procedure: Oral glucose tolerance test; Procedure: IV Glucose Tolerance Test
- Euglycemic Kidney Transplant Recipients (Active Comparator): Participants receiving a kidney transplant who have blood glucose level is within the normal range
  Interventions: Procedure: Oral glucose tolerance test; Procedure: IV Glucose Tolerance Test
- Euglycemic Healthy Control Participants (Active Comparator): Participants who do not receive either a pancreas or kidney transplant who have blood glucose level is within the normal range
  Interventions: Procedure: Oral glucose tolerance test; Procedure: IV Glucose Tolerance Test

INTERVENTIONS:
Procedure: Oral glucose tolerance test — test done over 2 hours
Procedure: IV Glucose Tolerance Test — Done over 4 hours

SUMMARY:
The purpose of this study is to understand how the pancreas functions after transplantation and particularly why high blood sugar levels develop. It will also analyze the effect of the medicines used to prevent rejection on blood sugar levels.

The hypothesis to be tested is that hyperglycemia more than six months after successful pancreas transplant results from a defect in insulin secretion, insulin resistance, or both.

DETAILED DESCRIPTION:
Type I diabetes mellitus (DM1) is an autoimmune disease characterized by destruction of the insulin-secreting beta cells. Insulin replacement has been the cornerstone of therapy for patients with DM1. However, pancreas transplantation, utilizing the whole pancreas as a means to replace the destroyed beta cells, has become a therapeutic alternative. The goal of pancreas transplantation is the establishment of long-term euglycemia, thereby preventing or allowing for the repair of end-organ complications.

Maintenance of the pancreas allograft over many years remains the goal in following pancreas transplant recipients over time. The onset of hyperglycemia less than one year after transplant is usually due to issues of surgical technique or acute rejection. However, the onset of hyperglycemia after one year of pancreas transplant is more problematic because the underlying causes are less clear and have been less well characterized. Currently, there is no protocol for definitively identifying the causes of hyperglycemia in pancreas transplant recipients over one year. This project will systematically characterize beta cell function and peripheral tissue response to insulin in patients who have received an earlier successful pancreas transplant who have developed hyperglycemia.

ELIGIBILITY:
Inclusion Criteria:

* Hyperglycemic pancreas transplant recipients:

  * ages 19-65
  * received a pancreas transplant ≥ 9 months previously
  * fasting glucose levels ≥ 126 mg/dl
  * hemoglobin A1C > 1% above normal
* Euglycemic pancreas transplant recipients:

  * ages 19-65
  * received a pancreas transplant ≥ 9 months previously
  * fasting glucose levels are < 126 mg/dl
  * normal HbA1C without taking any medications for the treatment of high blood sugars.
* Euglycemic Kidney Transplant Recipients:

  * ages 19-65
  * no prior diagnosis of diabetes
  * received a kidney transplant ≥ 9 months previously
  * showing continued function
* Euglycemic Healthy Control Subjects:

  * ages 19-65
  * no diabetes or renal disease

Exclusion Criteria:

* Hyperglycemic pancreas transplant recipients:

  * chronic illnesses that would decrease insulin sensitivity (
  * terminal illness
  * BMI > 30 kg/m2
  * serum creatinine > 2 mg/dl
  * hemoglobin < 10 g/dl
  * an episode of acute rejection with the preceding 3 months of entry.
* Euglycemic pancreas transplant recipients:

  * Exclusion criteria are the same as with hyperglycemic transplant patients.
  * no diagnosis of type 2 diabetes.
* Euglycemic Kidney Transplant Recipients:

  * Exclusion criteria are the same as for euglycemic pancreas transplant recipients above.
* Euglycemic Healthy Control Subjects:

  * chronic illnesses
  * medications known to affect glucose metabolism
  * a history of smoking
  * serum creatinine ≥ 1.5 mg/dl
  * BMI > 30 kg/m2.

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2000-11-01 (Actual); Primary Completion 2008-03-01 (Actual); Study Completion 2010-06-01 (Actual)

PRIMARY OUTCOMES:
Evaluate beta cell secretion | 9 months post-transplant or at time of participation for controls
  Evaluate beta cell secretion by oral glucose tolerance test (done over 2 hours) and IV Glucose Tolerance Test (done over 4 hours)
Evaluate insulin sensitivity/glucose effectiveness | 9 months post-transplant or at time of participation for controls
  Evaluate insulin sensitivity/glucose effectiveness by oral glucose tolerance test (done over 2 hours) and IV Glucose Tolerance Test (done over 4 hours)

CONTACTS AND LOCATIONS:
Overall Officials: James T Lane, MD, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Omaha, Nebraska, United States